CLINICAL TRIAL: NCT02057016
Title: Long-term Scheduled Therapy With Infliximab in Inflammatory Bowel Disease: a Single-centre Observational Pilot Study
Brief Title: Long-term Scheduled Therapy With Infliximab in Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Alessandro Armuzzi, MD PhD, Catholic University of the Sacred Heart
Other Study IDs: LTIT-090114
Record Dates: First submitted 2014-02-05; First posted 2014-02-06 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Crohn's Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary objective of this study is to evaluate sustained clinical remission (for the definition see below) in patients with inflammatory bowel disease receiving long-term (> 2 years) scheduled treatment with infliximab.

Secondary objectives include:

* to identify predictors of sustained clinical remission during long-term infliximab scheduled treatment
* to identify predictors of loose of response during infliximab scheduled maintenance treatment
* to identify predictors for maintaining clinical remission in patients who discontinue infliximab because of long-lasting steroid-free clinical remission
* to evaluate percentage of surgery during and after treatment (total follow-up)
* to evaluate safety of long-term infliximab scheduled treatment

List the clinical hypotheses

Infliximab is indicated and recommended in moderate to severe inflammatory bowel disease patients who not tolerate or are not responsive to conventional therapies. Most of randomized clinical trials about the use of infliximab in inflammatory bowel diseases are limited to 52 weeks and very few data come from some observational studies about results of prolonged (over one year) treatment with infliximab. No validated predictors of sustained clinical remission or loss of response are available so far. Moreover, few data are available about the hypothetical reduction of IBD related surgery in the "biological era".

In this proposal we suggest the following hypotheses:

* infliximab scheduled treatment may be efficacious in maintain long-term clinical remission;
* among clinical, laboratory and endoscopic data some predictors of sustained clinical remission during infliximab long-term scheduled treatment may be found;
* among clinical, laboratory and endoscopic data some predictors of loss of response during infliximab long-term scheduled treatment may be found;
* among clinical, laboratory and endoscopic data some predictors of sustained clinical remission after infliximab discontinuation because of long-lasting (> 6 months) steroid-free clinical remission may be found;
* maintenance of remission with infliximab may reduce rates of surgery over time;
* long-term scheduled treatment with infliximab may be safe and well tolerated. Results from this study may really help clinicians to make practical decisions in these particular clinical settings.

DETAILED DESCRIPTION:
Study design:

This is a retrospective observational "real life" single-centre study.

Materials and methods:

Medical records of all IBD patients who continued maintenance treatment with infliximab being in clinical remission after one year of scheduled therapy (standard induction and maintenance dose) will be considered eligible for this study.

Demographic, clinical, laboratory and endoscopic data and adverse events will be reported in a database. In particular, data available for each patient will concern:

* age,
* sex,
* smoker status,
* Montreal classification,
* disease duration,
* activity of disease,
* previous surgery,
* concomitant arthritis,
* concomitant corticosteroids,
* previous or concomitant immunosuppressives,
* eventual infliximab dose escalation,
* total number of infliximab infusions,
* reason of eventual infliximab discontinuation,
* time on infliximab therapy,
* total follow-up since the first infliximab infusion,
* IBD related surgeries,
* endoscopic data within the first year and beyond up to infliximab discontinuation time,
* laboratory data (C-reactive protein and hemoglobin levels),
* adverse events.

Clinical remission will be evaluated using the Harvey-Bradshaw Index (HBI) in Crohn's patients (HBI ≤ 4) and the partial Mayo score in UC patients (<2 with rectal bleeding subscore = 0).

Sustained clinical remission will be defined as a HBI ≤ 4 or partial Mayo score < 2 (with rectal bleeding = 0) after 54 weeks from baseline.

At the baseline of the study all patients should have already received one year of infliximab scheduled treatment and should be in clinical remission (as defined above).

Primary endpoint will be evaluated at week 54 from baseline (after 2 overall years of treatment) and then every year during the follow-up.

Secondary endpoints will be evaluated considering all available data at the end of follow-up.

Number of patients:

232 IBD (131 CD, 101 UC)

Procedures:

All IBD patients treated for at least one year with infliximab because of active luminal Crohn's disease and active ulcerative colitis will be included in this study.

Infliximab administration has been done according to SPC. Due to retrospective and observational pattern of the study, clinical management of patients depended on practice in our IBD unit. In particular, patients were clinically evaluated by visits at every infusion of infliximab. Also laboratory tests were periodically repeated (every two months).

No therapeutic changes were made in consideration of the present study. The indications to start infliximab treatment corresponded to those reported in international guidelines.

This study will be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki and will be consistent with International Conference on Harmonization Good Clinical Practice (ICH GCP), Good Epidemiological Practices(GEP) and applicable regulatory requirements taking into account that this is an observational, non-interventional trial.

Statistical analysis:

Data will be described using medians with interquartile range (IQR) for continuous data and percentages for discrete data.

Kaplan-Maier survival curves will be performed to reveal the variables that may influence primary and secondary endpoints.

To compare hazard rates in populations defined by one variate at a time, Cox proportional hazard analysis will, then, be performed with the aim to identify predictors of maintenance of remission while on IFX treatment and after IFX discontinuation, and predictors of loss of response during scheduled maintenance therapy with IFX.

Principal variables used for the statistical evaluation will include: sex, age at diagnosis, disease duration, smoking status, previous surgery, disease location, disease extension, concomitant arthritis, endoscopic activity (mucosal healing), CRP and hemoglobin levels, previous immunomodulators, concomitant immunomodulators, need for dose escalation.

ELIGIBILITY:
Inclusion Criteria:

* patients with inflammatory bowel disease receiving long-term (> 2 years) scheduled treatment with infliximab

Exclusion Criteria:

* patients with inflammatory bowel disease who received less than 2-year scheduled treatment with infliximab

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with inflammatory bowel disease receiving long-term (> 2 years) scheduled treatment with infliximab
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Efficacy outcome | 2 years
  Evaluation of sustained clinical remission in patients with inflammatory bowel disease receiving long-term (> 2 years) scheduled treatment with infliximab

SECONDARY OUTCOMES:
Efficacy outcome | 2 years
  Evaluation of predictors of sustained clinical remission during long-term infliximab scheduled treatment, predictors of loose of response during infliximab scheduled maintenance treatment and predictors for maintaining clinical remission in patients who discontinue infliximab because of long-lasting steroid-free clinical remission
Safety outcome: Evaluation of safety of long-term infliximab scheduled treatment. | 2 years
  Adverse events (AE) will be retrospectively reported in the database following this definition of terms.
  Per the International Conference on Harmonization (ICH), an AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product.
  Serious Adverse Event is any untoward medical occurrence or effect that at any dose: results in death, is life-threatening; requires hospitalization or prolongation of existing inpatients' hospitalization; results in persistent or significant disability or incapacity; and/or is a congenital anomaly or birth defect; is a cancer; is associated with an overdose; is another Important Medical Event.

OTHER OUTCOMES:
Surgery outcome | 2 years
  Evaluation of percentage of surgery during and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- IBD Unit, Complesso Integrato Columbus, Catholic University of the Sacred Heart, Rome, RM, Italy